CLINICAL TRIAL: NCT02542189
Title: High Sensitivity Cardiac Troponin T in Patients With Atrial Fibrillation Admitted to an Emergency Department (ED)
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Professor Hugo Katus, MD, PhD, FESC; FACC, University Hospital Heidelberg
Other Study IDs: S-377-2013
Record Dates: First submitted 2015-08-06; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to collect data on the prevalence and clinical significance of elevated cardiac troponin in a large registry of unselected patients with atrial fibrillation presenting to an emergency department.

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrillation in admission EKG or diagnosis of atrial fibrillation at admission.

Exclusion Criteria:

* no patients are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of approximately 3,500 consecutive patients presenting to the emergency department of the University Clinic Heidelberg between June 2009 and March 2013.
Sampling Method: Probability Sample
Enrollment: 3037 (Actual)
Dates: Start 2009-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
vascular and non-vascular death | up to 60 months
  Assessment via review of inpatient- and outpatient visit reports, patient phone calls, postal queries with standardised questionnaires, contact with primary care physicians and resident registration office inquiries.
nonfatal myocardial infarction | up to 60 months
  Assessment via review of inpatient- and outpatient visit reports, patient phone calls, postal queries with standardised questionnaires, contact with primary care physicians and resident registration office inquiries.
stroke/transitory ischemic attack (TIA) | up to 60 months
  Assessment via review of inpatient- and outpatient visit reports, patient phone calls, postal queries with standardised questionnaires, contact with primary care physicians and resident registration office inquiries.

REFERENCES:
- [Derived] Stoyanov KM, Giannitsis E, Biener M, Mueller-Hennessen M, Arens K, Katus HA, Vafaie M. Prognostic value of elevated high-sensitivity cardiac troponin T in patients admitted to an emergency department with atrial fibrillation. Europace. 2018 Apr 1;20(4):582-588. doi: 10.1093/europace/eux063. PMID 28460039